CLINICAL TRIAL: NCT00274794
Title: A Prospective Randomized Trial of VP-16 Plus G-CSF Plus Rituximab vs VP-16 Plus G-CSF Alone for Peripheral Blood Progenitor Cell Mobilization Prior to Autologous Stem Cell Transplantation for B Cell Lymphoid Malignancies
Brief Title: VP and G-CSF With or Without Rituximab in Autologous Peripheral Stem Cell Transplant For NHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Brian Bolwell, MD, Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE-CCF-3600; P30CA043703 (NIH); CASE-CCF-3600; CASE-CCF-0467
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Lymphoma
Keywords: noncontiguous stage II adult Burkitt lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; recurrent adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituxan + Etoposide + G-CSF (Other)
  Interventions: Biological: filgrastim; Biological: rituximab
- Etoposide + G-CSF (Other)
  Interventions: Biological: filgrastim

INTERVENTIONS:
Biological: filgrastim — 10mcg/kg/d subcutaneously, beginning 48 hours after completion of Etoposide
Biological: rituximab — 375 mg/m2, IV, Once per week for 3 weeks.
  Arms: Rituxan + Etoposide + G-CSF

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as busulfan, etoposide, and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving colony-stimulating factors, such as G-CSF, monoclonal antibodies, such as rituximab, or chemotherapy, such as etoposide, helps stem cells move from the bone marrow to the blood so they can be collected and stored until transplant. Giving etoposide and G-CSF together with rituximab before a peripheral stem cell transplant may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: This randomized clinical trial is studying how well giving etoposide and G-CSF with or without rituximab works in treating patients who are undergoing an autologous peripheral stem cell transplant for B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether mobilization with etoposide and filgrastim (G-CSF) with or without rituximab influences CD34+ cell yield in patients undergoing autologous peripheral blood stem cell transplantation for B-cell non-Hodgkin's lymphoma.
* Determine the acute toxicity of rituximab in combination with etoposide and G-CSF for peripheral blood stem cell mobilization in these patients.

OUTLINE: This is a randomized study.

* Stem cell mobilization: Patients are randomized to 1 of 2 mobilization arms.

  * Arm I: Patients receive rituximab IV over 4 hours on days 1, 8, and 15. Patients also receive etoposide IV over 4 hours on day 15 and filgrastim (G-CSF) subcutaneously (SC) beginning on day 17 and continuing until approximately day 25. Patients then undergo apheresis over 5 days or until an adequate amount of stem cells are collected. After stem cell collection is completed, patients proceed to the preparative regimen.
  * Arm II: Patients receive etoposide IV over 4 hours on day 1 and G-CSF SC beginning on day 3 and continuing until approximately day 11. Patients then undergo apheresis over 5 days or until an adequate amount of stem cells are collected. After stem cell collection is completed, patients proceed to the preparative regimen.
* Preparative regimen: Patients receive oral busulfan once daily on days -8 to -4, etoposide IV over 4 hours on day -4, and cyclophosphamide IV over 2 hours on days -3 and -2.
* Autologous peripheral blood stem cell transplantation (PBSCT): Patients undergo autologous PBSCT on day 0. Beginning on day 5, patients receive G-CSF SC or IV once daily until blood counts recover.

After completion study treatment, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients with B-cell malignancies who are appropriate candidates for high-dose chemotherapy and autologous stem cell transplantation and meet 1 of the following criteria:

  * Relapsed or refractory B-cell non-Hodgkin's Lymphoma (NHL)
  * Patients with B-cell NHL in first remission and who have significant risk for later relapse
  * Patients with other B-cell malignancies otherwise eligible for autologous stem cell transplantation

PATIENT CHARACTERISTICS:

* Life expectancy at least 2 months
* Cardiac ejection fraction ≥ 45%
* DLCO ≥ 45%
* Creatinine < 2.0 mg/dL
* Bilirubin < 2.0 mg/dL
* AST < 2 times normal
* Platelet count ≥ 50,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Absolute lymphocyte count ≤ 10,000/mm^3
* HIV negative
* No severe medical or psychiatric illnesses
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* More than 8 weeks since prior rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2000-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Correlate CD34+ cell yields with the addition of rituximab | At least two weeks prior to transplant
Acute toxicity of rituximab, etoposide, and filgrastim (G-CSF) | 100 days post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Bolwell, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio, United States

REFERENCES:
- [Result] Copelan E, Pohlman B, Rybicki L, Kalaycio M, Sobecks R, Andresen S, Dean R, Koo A, Chan J, Sweetenham J, Bolwell B. A randomized trial of etoposide and G-CSF with or without rituximab for PBSC mobilization in B-cell non-Hodgkin's lymphoma. Bone Marrow Transplant. 2009 Jan;43(2):101-5. doi: 10.1038/bmt.2008.306. Epub 2008 Sep 15. PMID 18794865